CLINICAL TRIAL: NCT06575816
Title: Effect of Augmented Reality on Pain, Anxiety and Fear During Blood Collection in Children: Randomized Controlled Study
Brief Title: Effect of Augmented Reality on Pain, Anxiety, and Fear in Children During Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Emine Zahide Özdemir, Assistant Professor Doctor, PhD, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DokuzEU-2024
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-08

CONDITIONS: Pain; Fear; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group, intervention group (Active Comparator): This group will receive the standard blood collection procedure without any augmented reality video intervention. Pain, anxiety, and fear levels will be assessed using standardized scales after the procedure.
  This group will receive the augmented reality video intervention during the blood collection procedure. The intervention consists of children watching AR videos designed to distract and comfort them during the blood draw. Pain, anxiety, and fear levels will be measured using standardized scales immediately after the procedure.
  Interventions: Behavioral: Augmented Reality Video Intervention
- Control group (No Intervention): This group will receive the standard blood collection procedure without any augmented reality video intervention. Pain, anxiety, and fear levels will be assessed using standardized scales after the procedure.
- intervention group (Experimental): This group will receive the augmented reality video intervention during the blood collection procedure. The intervention consists of children watching AR videos designed to distract and comfort them during the blood draw. Pain, anxiety, and fear levels will be measured using standardized scales immediately after the procedure.
  Interventions: Behavioral: Augmented Reality Video Intervention

INTERVENTIONS:
Behavioral: Augmented Reality Video Intervention — This intervention involves a video intervention using augmented reality (AR) technology to reduce the pain, anxiety and fear children experience during the blood collection process. During the intervention, children watch AR videos to distract and relax them from the blood collection process. These videos are equipped with a variety of entertaining and engaging content and aim to reduce children's psychological stress.
  Arms: Control group, intervention group; intervention group

SUMMARY:
In recent years, technological advances have enabled the development of innovative intervention methods in healthcare. This study aims to examine the effect of augmented reality (AR) technology on pain, anxiety and fear in children during pediatric blood collection procedures. The study is based on a randomized controlled design. Participants were randomized into two groups, the group receiving AR intervention and the control group receiving standard care. Pain, anxiety and fear levels will be assessed with pre and post intervention measurements.

ELIGIBILITY:
Inclusion Criteria:

* Both parent and child voluntarily agree to participate in the study
* No language barrier

Exclusion Criteria:

* Parents or children who refused to participate in the study
* Problems with looking at the screen

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Pain Level | Five minutes before and 5 minutes after blood collection
  Children's pain levels will be measured using a standardized pain scale, such as the Wong-Baker Pain Rating Scale, immediately after the blood collection procedure.The scale can be scored from a minimum of 0 to a maximum of 10. As the score increases, pain increases.

SECONDARY OUTCOMES:
Fear Level | Five minutes before and 5 minutes after blood collection
  Children's fear levels will be evaluated using a fear assessment tool, such as the Children's Fear Scale, before and after the blood collection procedure.
  The scale can be scored from a minimum of 0 to a maximum of 4. As the score increases, fear increases.

OTHER OUTCOMES:
Anxiety Level | Five minutes before and 5 minutes after blood collection
  Children's anxiety levels will be assessed using the State-Trait Anxiety Inventory for Children before, during, and after the blood collection procedure.The scale can be scored from a minimum of 1 to a maximum of 10. As the score increases, Anxiety increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Zahide Özdemir, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No